CLINICAL TRIAL: NCT01642420
Title: Quantitative Electroencephalography, Cerebrospinal Fluid Biomarkers, Linear CT Analyses and Timed Up and GO Dual Task as Diagnostic Tools in Dementia and Their Ability to Predict Disease Progression.
Brief Title: Non-expensive and Widely Available Tests as Diagnostic Tools in Dementia and Their Ability to Predict Disease Progression
Acronym: DEMPROG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zealand University Hospital (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Malene Schjønning Nielsen, MD, PhD student, Zealand University Hospital
Other Study IDs: DEMPROG 2012
Record Dates: First submitted 2012-04-13; First posted 2012-07-17 (Estimated); Last update posted 2012-09-13 (Estimated); Status verified 2012-09

CONDITIONS: Alzheimers Disease; Mild Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Cerebrospinalfluid (CSF) CSF is analysed to find Alzheimer Disease biomarkers
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Mild cognitive impairment: Patients diagnosed with mild cognitive impairment
- Alzheimers disease: Patients diagnosed with mild Alzheimers disease
- Healthy control persons: Age matched healthy persons

SUMMARY:
Alzheimers disease (AD) is the most common course of cognitive decline and thereby the course of more than half of all cases of dementia. A proper AD diagnosis is rested on a number of examinations and tests, which combined can make AD diagnosis likely. But no single test or examination can unambiguous determine whether the patient has AD or not. Comparatively no examination or test can with accuracy predict whether a healthy person or a person with only mild cognitive (MCI)impairment in time will evolve AD.

Quantitative Electroencephalography (qEEG), cerebrospinal fluid (CSF) biomarkers, linear CT analyses and Timed Up and Go - Dual Task (TUG-DT) are relatively inexpensive and and widely available diagnostic methods, which have the potential to diagnose AD at an early stage in a reliable accurate way. But they also have the potential to predict which patients diagnosed with MCI have particular risk of developing dementia.

The purpose of the study is to investigate the relations between qEEG, CSF biomarkers, CT analyses and TUG-DT outcome and clinical features in healthy persons as well as patients with MCI and AD Furthermore to investigate whether qEEG or CSF biomarkers can predict which patients with MCI will in time evolve AD.

ELIGIBILITY:
Inclusion Criteria:

For patients:

* age 50 to 90
* diagnosed with MCI or AD
* cerebrospinal fluid examination and EEG performed at baseline

For control persons:

* age 50 to 90
* MMSE score equal or above 26
* ACE score equal or above 85
* Normal physical examination, including normal blood samples, CT of cerebrum and EEG examination

Exclusion Criteria:

* Pregnant or breastfeeding
* psychiatric disease, former depression is allowed if antidepressive treatment has been initiated of a leat 3 months duration
* Neurologic or somatic disease, including former severe head trauma or neuroinfection
* Antipsychotic treatment
* Former severe abuse of alcohol, medication or drugs
* ECT treatment or anaesthesia within the last 3 months
* no closely related person to assist the patient

Additionally exclusion criteria for healthy control persons:

* meet the diagnostic criteria for MCI or AD

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with MCI and AD will be recruitted among consectutively refered patients in a memory clinic. Participation is voluntary Healthy control persons will be recuitted by posters and notices
Sampling Method: Non-Probability Sample
Enrollment: 115 (Estimated)
Dates: Start 2012-04; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Conversion from Mild Cognitive Impairment to Alzheimers disease | Every year in totally of 3 years
  The primary outcome measure is progression of clinical symptoms to an extent where the formal NINCDS-ADRDA criteria for dementia is meet. The progression is based upon clinical symptoms as well as explorative determinants in form of clinical tests, CSF analysis and qEEG analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Malene S Nielsen, MD, Principal Investigator — Roskilde Hospital, Department of Neurology
Locations (1):
- Neurologisk Afd, Roskilde Sygehus, Roskilde, Denmark